CLINICAL TRIAL: NCT07224854
Title: A Model of Epigenetic Biomarkers Based on cfDNA 5mC/5hmC for Early Detection of Colorectal Cancer
Brief Title: Epigenetic Signature for CRC Early Detection
Acronym: epiCED
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/epiCED
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (Diagnosis); Non-cancer Controls; DNA Methylation; Cell Free DNA; Early Detection of Cancer
Keywords: noninvasive screening; circulating cfDNA; 5mC; 5hmC; epigenetic biomarkers; machine learning; colorectal cancer; early detection
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRC: Adult patients with confirmed colorectal cancer from international centers.
- Control: Non-cancer individuals, including healthy volunteers or patients with benign gastrointestinal conditions.

SUMMARY:
The epiCED is a noninvasive blood-based assay designed for early detection of colorectal cancer (CRC) using circulating cell-free DNA (cfDNA) 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) epigenetic markers. This study leverages retrospective, multi-center cohorts of CRC patients and non-cancer controls to discover and validate a robust cfDNA methylation signature. Small-scale sequencing and machine learning-based modeling will be applied to identify a minimal panel of methylation markers that can accurately discriminate CRC from non-cancer individuals, including early-stage disease. The ultimate goal is to develop a clinically practical, noninvasive screening tool that enables population-level early detection and improves patient outcomes.

DETAILED DESCRIPTION:
The epiCED is a noninvasive, blood-based approach aimed at early detection of colorectal cancer (CRC) using circulating cell-free DNA (cfDNA) 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) epigenetic markers. Early detection of CRC is critical for improving patient outcomes, but current diagnostic tools-including colonoscopy, CT, and MRI-are either invasive, costly, or insufficiently sensitive for early-stage disease, limiting their use for population-wide screening.

This study will utilize retrospective, multi-center cohorts comprising adult participants (≥18 years) with confirmed CRC and non-cancer controls, including healthy volunteers and individuals with benign gastrointestinal conditions. Blood samples will be subjected to cfDNA extraction and small-scale epigenetic sequencing to profile 5mC and 5hmC patterns.

During the discovery phase, differential methylation analysis and machine learning-based feature selection will be applied to identify a minimal set of cfDNA methylation markers that optimally discriminate CRC from non-cancer individuals. In the training and validation phase, the identified signature will be evaluated across independent international multi-center cohorts to ensure reproducibility, robustness, and early-stage detection performance.

The primary objectives are to:

* Develop a cfDNA methylation panel capable of accurately distinguishing CRC patients from non-cancer controls.
* Validate the panel's ability to detect early-stage CRC.
* Secondary objectives include evaluating the association of the methylation signature with clinical parameters, tumor stage, and demographic factors. By integrating high-resolution cfDNA methylation profiling with advanced computational modeling, epiCED aims to provide a scalable, cost-effective, and clinically practical tool for noninvasive early detection of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years at the time of sample collection.
* Patients with confirmed CRC or non-cancer controls.
* Availability of retrospective blood samples collected according to institutional protocols.
* Willingness to allow use of de-identified clinical and demographic data.

Exclusion Criteria:

* Concurrent malignancies outside the gastrointestinal tract (unless in complete remission ≥5 years).
* Samples with insufficient volume or poor cfDNA quality.
* Recent chemotherapy, radiotherapy, or major surgery within 4 weeks prior to blood collection (if prospective samples).
* Any condition precluding reliable sample analysis or participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective, international multi-center cohort of adults (≥18 years), including CRC patients and non-cancer controls. Blood samples and corresponding de-identified clinical data are available for discovery, model training, and multi-center validation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for detecting colorectal cancer | Baseline (pre-treatment blood sample collection)
  Proportion of true positive CRC cases correctly identified by the cfDNA methylation panel.

SECONDARY OUTCOMES:
Specificity for detecting colorectal cancer | Frame: Baseline (pre-treatment blood sample collection)
  Proportion of true negative (non-cancer) individuals correctly classified by the cfDNA methylation panel.
Area Under the Receiver Operating Characteristic Curve (AUROC) | Baseline (pre-treatment blood sample collection)
  AUROC of the cfDNA methylation panel for distinguishing CRC patients from non-cancer controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Nat Medical Ctr, Monrovia, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goddard KAB, Feuer EJ, Mandelblatt JS, Meza R, Holford TR, Jeon J, Lansdorp-Vogelaar I, Gulati R, Stout NK, Howlader N, Knudsen AB, Miller D, Caswell-Jin JL, Schechter CB, Etzioni R, Trentham-Dietz A, Kurian AW, Plevritis SK, Hampton JM, Stein S, Sun LP, Umar A, Castle PE. Estimation of Cancer Deaths Averted From Prevention, Screening, and Treatment Efforts, 1975-2020. JAMA Oncol. 2025 Feb 1;11(2):162-167. doi: 10.1001/jamaoncol.2024.5381. PMID 39636625
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751